CLINICAL TRIAL: NCT03986047
Title: Effect of Thermal Therapy in Combination With Exercises to Relieve Acute Low Back Pain
Brief Title: Effect of Thermal Therapy and Exercises on Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Quebec Pain Research Network (Other)
Responsible Party: Principal Investigator, Hugo Massé-Alarie, Adjunct professor, Rehabilitation Department, Faculty of Medicine, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Heat and exercises for ALBP
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
Keywords: Thermal therapy; Exercises; Pain; Disability; Acute pain
MeSH Terms: conditions — Low Back Pain; Motor Activity; Pain; Acute Pain | interventions — Exercise; Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized control trial, as following :
  * Baseline evaluation
  * Randomized assignment to one of 3 intervention groups (Thermal + Exercises, Thermal alone, and Control)
  * Post-intervention assessment (current pain)
  * 1-week home-based intervention
  * Reassessment at 1 week, 1 month, 3 months, 6 months
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessor is blinded to participant's intervention allocation. Participants are blinded to the nature of interventions given in the other arms' groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermal care (Experimental): Participants will be asked to wear a heat wrap over the lower lumbar spine, during the day for 8 hours on 7 consecutive days. The Thermal care group will also receive education by a physiotherapist on acute low back pain management.
  Interventions: Device: Thermal care; Behavioral: Education for the management of acute low back pain
- Thermal care + exercises (Experimental): In addition to heat wrap and pain management education as for Thermal care group, participants of this group will be asked to perform exercises at home over 7 days, targeted on functional capacity, lumbar mobility, and slight contraction of trunk muscle (posture and/or cognitive).
  Interventions: Device: Thermal care; Other: Exercises; Behavioral: Education for the management of acute low back pain
- Control (Sham Comparator): Participants in the control group will receive the same education program as those of the two other groups. A sham non-heating wrap will be used to control for potential supportive and sensory influence of the heat wrap.
  Interventions: Device: Sham; Behavioral: Education for the management of acute low back pain

INTERVENTIONS:
Device: Thermal care — Wearing of a light elastic lower back heating wrap, which heats up to 40°C within 30 minutes and maintains this temperature continuously for 8 hours. Heat wrap will be worn during the day for 8 hours on 7 consecutive days.
  Other Names: ThermaCare® Back Pain Therapy HeatWraps, by Pfizer
  Arms: Thermal care; Thermal care + exercises
Other: Exercises — In addition of exercises performed with the physiotherapist at the first session, exercises will be performed at home five times over the next 7 days, for approximately 30 minutes each performing day. Three different categories of exercises will be given: 1) Functional activities exposure (sitting, sit-to-stand, lifting, bending, etc.); 2) cognitive contraction of trunk muscles and basic trunk motor control exercises; 3) mobility of the lumbar spine and preferential direction of movement. Exercises will be chosen and adapted for each participant by a physiotherapist, in function of pain presentation and intensity, and response to exercises.
  Arms: Thermal care + exercises
Device: Sham — The same lower back wrap as the Thermal care group will be used, but cooled down to room temperature (opened in advance). The wrap will be worn following the same parameters (duration, frequency) than the Thermal care group.
  Arms: Control
Behavioral: Education for the management of acute low back pain — Participants will receive education on the management of acute low back pain by a physiotherapist . The main topics addressed will be patient reassurance, staying active, avoiding bed rest, activity modification, and sitting and bed postures/transfer. Participants will received a document that details advices covered during the session and the physiotherapist will answer any questions.

SUMMARY:
Low back pain (LBP) ranks among the first diseases in term of years lived with disability. The latest Clinical Guideline from the American College of Physicians for acute LBP recommends to select "nonpharmacologic treatment with superficial heat, massage, acupuncture or spinal manipulation". The application of superficial heat ("thermal therapy") may provide enough pain relief in the acute phase to remain active, which is recommended to prevent the development of chronicity. However, no studies have tested if the combination of heat and exercises provide additional benefit on short, middle and long-term follow-up in people with acute LBP.

Hence, the main objective of this study is to determine the immediate, short-, middle- and long-term effect of continuous low-level thermal therapy in combination or not with exercises on pain, disability, and physical activity level in people with acute LBP.

Project hypothesis : The Thermal care + Exercises group will show greater improvement in pain, disability and physical activity level than both Thermal care and Control groups for immediate, short-, middle- and long-term follow-ups.

Sixty individuals with acute LBP will be recruited. This study will include six assessments over 6 months. At the baseline evaluation, participants will complete questionnaires on symptoms, disability, pain-related fear and self-efficacy. Afterwards, participants will be randomly assigned to one of three intervention programs: 1) Thermal care group, 2) Exercises + Thermal care group, and 3) Control group. They will immediately meet a physical therapist to review and perform their assigned program.

Participants will then take part in their assigned 7-day intervention program, during which they will wear a fitness wristband to track physical activity level. Finally, the same outcomes will be reassessed to determine the effect of intervention at 1 week, 1 month, 3 months and 6 months after baseline.

DETAILED DESCRIPTION:
Low back pain (LBP) ranks among the first diseases in term of years lived with disability, which is mostly explained by the development of recurrent or chronic pain. A systematic review observed that 62% of patients still have pain 12 months after onset (recurrent and chronic) while another estimated that between 2% and 34% of acute cases will develop chronic LBP. These rates highlight the need to identify the best therapeutic approaches at the acute stage to prevent transition to chronicity and high recurrence. The latest Clinical Guideline from the American College of Physicians for acute LBP recommends to select "nonpharmacologic treatment with superficial heat, massage, acupuncture or spinal manipulation". The application of superficial heat ("thermal therapy") presented the strongest evidence (moderate) for short-term reduction in pain. Four randomized controlled trials (RCT) that tested the effect of a wearable heatwrap (the most studied form of thermal therapy in acute LBP) reported a reduction in pain and disability up to 2 days after cessation of the intervention: an effect superior to Ibuprofen, Acetaminophen or oral placebo. Heatwrap may provide enough pain relief in the acute phase to remain active, which is recommended to prevent the development of chronicity. One RCT showed that the addition of a heatwrap to exercise provided greater short-term improvement in pain/disability than exercise alone. Although some authors suggest that an increase in physical activity level may explain such an effect, this assumption has not been tested yet.

Hence, the main objective of this RCT is to determine the immediate, short-, middle- and long-term effect of continuous low-level thermal therapy in combination or not with exercises on pain, disability, and physical activity level in people with acute LBP.

Project hypothesis : The Thermal care + Exercises group will show greater improvement in pain, disability and physical activity level than both Thermal care and Control groups for immediate, short-, middle- and long-term follow-ups.

Participants: Individuals with acute LBP will be included according to the mentioned inclusion/exclusion criteria. They will be recruited from medical and through the electronic mailing list of Université Laval (> 52,000 individuals). The list of participants of the Quebec Low Back Pain Study (QLBPS Core Dataset, funded by the QPRN) will also be used - all participants in the Quebec City area recruited for the QLBPS Core Dataset will be referred for the present project.

Study Design: This study will include six assessments over 6 months : baseline pre, 1-hour post, 1 week, 1 month, 3 months, 6 months. At the baseline evaluation (baseline pre), participants will complete self-administered questionnaires on symptoms and disability (Numerical scale for pain, Oswestry Disability Index - ODI, Global Rating of Change - GRC), on pain-related fear (Tampa Scale of Kinesiophobia - TSK) and on pain-related self-efficacy (Chronic Disease Self-Efficacy Scale short version - CDSES-6). Finally, participants will be randomly assigned to one of three intervention programs: 1) Thermal care group, 2) Thermal care + Exercises group, and 3) Control group. Immediately after group assignment (same session), participants will meet a physical therapist (PT) to review their assigned program (60-minutes meeting), during which a ThermaCare® Heat wrap or a sham wrap will be applied by the PT. In Thermal Care + Exercises group, an exercise program will be taught by the PT then performed by participants. General advices on the management of acute LBP will be given to all participants. Thereafter, the immediate effect of thermal therapy on pain will be evaluated (1-hour post-intervention assesment).

After the baseline evaluation and PT session, participants will perform their assigned 7-day intervention program. Every day, they will complete a logbook related to their pain level during the previous day and to their adherence to their program. In addition, participants will wear a fitness wristband to track physical activity level for 7 days (number of steps per day). Then, pain, ODI, GRC, TSK and CDSES-6 will be assessed at 1 week, 1 month, 3 months and 6 months after baseline to determine short-, middle-, and long-term effect of interventions.

Randomisation: a list will be generated using a computer random number generator by an independent research assistant (allocation concealed in sealed and opaque envelopes).

Sample size & Statistical analyses: Based on sample size calculation, calculated for the primary outcome (ODI) and previous data from the project investigators group (n=50 with acute LBP), 20 participants are required per group (G*Power 3.1.7; effect size: 0.80, α = 0.05, β = 0.80, mean baseline ODI of 44.0 +/- 13.5, lost at follow-up = 10%). Thus, 60 participants with acute LBP will be recruited.

To determine the effect of interventions, two-way ANOVA (Group x Time) will be performed (after confirming normality and homogeneity of variance). Bonferroni adjustments for multiple comparisons will be used (posthoc), and effect sizes will be reported (η2).

ELIGIBILITY:
Inclusion Criteria:

* to be suffering from low back pain (LBP) for a period of less than 6 weeks (with or without leg pain) that had limited one's activities or changed the daily routine for more than a day,
* to have been pain free for at least 3 months before the onset of the current LBP episode.

Exclusion Criteria:

* "red flag" signs that may suggest serious spinal pathology,
* history of spinal surgery,
* obvious lower limb radiculopathy
* fibromyalgia
* rheumatoid arthritis
* important skin lesion in the lumbar area
* alteration of cutaneous sensations or temperature perception
* being pregnant of trying to become

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in functional limitations and symptoms measured with the Oswestry Disability Index (ODI) version 2.1 | Change from baseline at 1-week, 1-month, 3-month and 6-month follow-up
  A list of ten items to assess symptoms (low back pain) and the functional disability it has caused in 9 different areas of everyday life. Score ranges from 0 to 100.

SECONDARY OUTCOMES:
Immediate change in current pain intensity after a 1-hour intervention with a numerical rating scale. | Change from baseline to 1 hour (after a 1-hour intervention)
  11-points rating scale (0 to 10), ranging from ''No pain'' to ''Worst pain imaginable''
Change in ''average pain intensity during the last 24 hours'' at 1 week measured with a numerical rating scale. | Change between baseline and after the 1-week intervention
  11-points rating scale (0 to 10), ranging from ''No pain'' to ''Worst pain imaginable''
Change in ''average pain intensity during the last 7 days'' measured with a numerical rating scale. | Change from baseline at 1-month, 3-month and 6-month follow-ups
  11-points rating scale (0 to 10), ranging from ''No pain'' to ''Worst pain imaginable''
Change in pain-related fear measured with Tampa Scale of kinesiophobia (TSK-11). | Change from baseline at 1-week, 1-month, 3-month and 6-month follow-up
  11-item version of the TSK questionnaire that measures problematic beliefs and behaviours associated with pain, focusing on beliefs that pain is damaging and that painful movements should be avoided. Each item is rated on a 4-point Likert scale (1=strongly disagree, 4=strongly agree). The total score ranges from 11 to 44 points, and higher scores signify greater fear of re-injury due to movement.
Change in self-efficacy measured with the Chronic Disease Self-Efficacy Scale - Short-Version (CDSES-6) | Change from baseline at 1-week, 1-month, 3-month and 6-month follow-up
  6-item version of the CDSES-33 questionnaire which measures the self-efficacy to perform behaviors and to achieve outcomes among those with chronic diseases (also validated with chronic pain for French Canadian population). Each item is measured using a numerical scale ranging from 1 (not at all confident) to 10 (totally confident). The total score is obtained by calculating the mean of the 6 items and ranges from 1 to 10. Higher scores indicate higher self-efficacy.
Change in physical activity level at 1 week, assessed by the number of steps walked per day. | Difference between groups at 1 week
  Measured with a fitness wristband
Global Rating of Change | Collected at 1-week, 1-month, 3-month and 6-month follow-up
  A single-item question that asks whether and to what extent the patient perceive change in his global lower back pain condition has occurred, since the initial evaluation, on a 15-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Massé-Alarie, Principal Investigator — Laval University, Quebec City
Locations (1):
- Centre interdisciplinaire de recherche en réadaptation et intégration sociale (CIRRIS), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cote-Picard C, Tittley J, Mailloux C, Perreault K, Mercier C, Dionne CE, Roy JS, Masse-Alarie H. Effect of thermal therapy and exercises on acute low back pain: a protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2020 Dec 5;21(1):814. doi: 10.1186/s12891-020-03829-7. PMID 33278897